CLINICAL TRIAL: NCT03556228
Title: A Phase 1/2 Open-Label, Multiple-Dose, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of VMD-928 as Monotherapy and in Combination With Pembrolizumab in Subjects With Solid Tumors or Lymphoma
Brief Title: VMD-928 Monotherapy and in Combination With Pembrolizumab to Treat TrkA Overexpression Driven Solid Tumors or Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VM Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VMO-01C
Record Dates: First submitted 2018-04-29; First posted 2018-06-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Carcinoma; Adenoid Cystic Carcinoma; Lung Cancer; Non-Small Cell Lung Cancer; Pancreatic Cancer; Mesothelioma; Esophageal Cancer; Any Solid Tumors Progressed After a Prior Immunotherapy; Head and Neck Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma HNSCC; Salivary Gland Carcinomas; Head and Neck Cancers - Salivary Gland; Head and Neck Cancers - Nasopharyngeal; Head and Neck Cancers - Throat; Small Cell Lung Cancer ( SCLC ); Lung Cancer (Locally Advanced or Metastatic); Head and Neck Cancers - Tonsils; Head and Neck Cancers Hypopharynx; Head and Neck Cancers Larynx; Head and Neck Cancers Lip; Head and Neck Cancers Nasopharynx; Head and Neck Cancers Oral Cavity; Head and Neck Cancers; Head and Neck Cancers Oropharynx; Head and Neck Cancers Trachea
Keywords: TrkA; NTRK1; Head and Neck Carcinoma; Adenoid Cystic Carcinoma; Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Mesothelioma; Pancreatic; Progression after anti PD-1/PD-L1 immunotherapy; Progressed after an immunotherapy; Esophageal; SCLC; ACC; HNSCC; Head and Neck Cancers; HNC; Salivary Gland Carcinoma; Nasopharyngeal; Throat; Tonsils; Hypopharynx; Larynx; Oral Cavity; Oropharynx; Trachea
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Mesothelioma; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Neoplasm Metastasis; Head and Neck Neoplasms; Salivary Gland Neoplasms; Laryngeal Diseases; Tracheal Diseases | interventions — Tablets; pembrolizumab; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: Tablet formulation and in Combination with Pembrolizumab:
  * Dose Escalation (Phase 1)
  * Cohort Expansion with RP2D (Phase 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VMD-928 monotherapy (Experimental): VMD-928 tablet monotherapy
  Interventions: Drug: VMD-928 100 mg Tablet
- Combination Therapy (Experimental): VMD-928 tablet in combination with fixed dose of pembrolizumab 200 mg once-very-21-day (per cycle)
  Interventions: Drug: VMD-928 Tablet and Pembrolizumab (200 mg)

INTERVENTIONS:
Drug: VMD-928 100 mg Tablet — Taken orally once daily for 21 days per 21-day cycle
  Other Names: Monotherapy
  Arms: VMD-928 monotherapy
Drug: VMD-928 Tablet and Pembrolizumab (200 mg) — VMD-928 tablet (oral) starting at 300 mg daily for 21 days of 21-day cycle. Pemprolizumab at fixed intravenous dose of 200 mg once-every-21 days (per cycle) for max. 6 cycles.
  Other Names: Combination therapy
  Arms: Combination Therapy

SUMMARY:
This is a multicenter, open-label, Phase 1/2 study of orally administered VMD-928 monotherapy and in combination with pembrolizumab in adult subjects with advanced solid tumors or lymphoma that have progressed or are non responsive to available therapies and for which no standard or available curative therapy exists

DETAILED DESCRIPTION:
This is an open-label, dose-escalation (Phase 1) and expansion (Phase 2) multi-center study conducted in five parts to identify the safe and pharmacologically active doses (MTD and/orRP2D) and regimen for oral VMD-928 monotherapy and in combination with a PD-1 inhibitor, pembrolizumab in cancer patients. An immunohistochemistry (IHC) assay specific for detecting TrkA protein in tumor tissue samples has been validated and is being used to detect TrkA protein expressions in patient tumor tissue samples at Pre-screening. The study is currently focusing on the top 5 solid tumor with the highest TrkA protein overexpression are: Head and Neck Cancers (HNC), Esophageal cancer, Lung cancers, Mesothelioma, and Pancreatic Cancer.

ELIGIBILITY:
Key Inclusion Criteria:

#. Histologically or cytologically confirmed diagnosis of any type of solid tumor malignancy or lymphoma:

Phase 1 Dose Escalation only: Subjects with

(A) any advanced solid tumors of

1. Head and Neck Cancers ("HNC") (of any types),
2. Esophageal cancer,
3. Lung cancers (of any types),
4. Mesothelioma,
5. Pancreatic cancers,

Or,

(B) any NTRK1 gene fusion positive ("NTRK1+") solid tumors or lymphomas, that is relapsed, refractory or intolerant (R/R/I) to standard of care (SOC) and for which there is no approved or curative therapy. Additionally, patients must not be candidates for or have exhausted regimens known to provide clinical benefit, including hematopoietic stem cell transplantation in lymphoma patients if they are deemed transplant eligible.

Phase 2 Monotherapy and Combination with Pembrolizumab only:

Subjects must have

1. TrkA-driven HNC, Esophageal, Lung, Mesothelioma, Pancreatic cancers; or,
2. any NTRK1+ solid tumors or lymphoma*, that is R/R/I to SOC.

Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0 or 1.
* Able to swallow and retain oral medication.
* Subjects must either have available archival tumor tissue samples, or consent to tumor tissue sampling prior to the first dose.
* Adequate organ system function as defined as follows:

  1. Absolute neutrophil count ≥1.5x10^9/L
  2. Hemoglobin ≥9g/dL
  3. Platelets ≥100x10^9/L
  4. PT/INR, PTT ≤1.5xULN
  5. Total bilirubin ≤1.5x ULN
  6. AST, ALT ≤2.5xULN
  7. Creatinine ≤1.2xULN for age, weight
  8. Calculated creatinine clearance or 24h urine creatinine clearance ≥60mL/min

Key Exclusion Criteria:

* Received chemotherapy having delayed toxicity within the last 14 days (six weeks for prior nitrosourea or mitomycin C).
* Received anticancer therapy with radiation, immunotherapy, and a biologic, surgery and/or tumor embolization within the past 2 weeks.
* Received an investigational anticancer drug within 14 days or 5 half-lives of the investigational agent, whichever is longer, prior to the first dose of VMD-928. Any exceptions to the above must be approved by the Sponsor Medical Monitor.
* Unresolved toxicity from previous anticancer therapy &gt; CTCAE Grade 1 (except alopecia or anemia) unless agreed to by both the Sponsor Medical Monitor and the Investigator.
* Known active infections including HIV disease.
* Currently pregnant, nursing, or planning to become pregnant during the course of the study.
* QTcF interval ≥ 480 msec.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks.
* Unstable or uncompensated respiratory, hepatic, renal, or cardiac disease that would compromise the patient's safety or interfere with assessment of the drug.
* Psychological, familial, sociological, geographical, or other concurrent conditions that would interfere with safety evaluation, limit the patient's ability to follow the procedures in the protocol or otherwise jeopardize compliance with the protocol. Patients with uncontrolled major depression, bipolar disorder, or severe anxiety disorder are excluded.
* Patient has had or is currently having other malignant tumors within 3 years.
* Patients have multiple factors that affect their oral medication.
* Patients have long-term unhealed wounds or fractures.
* Patients have uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage.
* Patients are taking the following drugs and can't stop them during the study:

  * Tylenol or medicine containing acetaminophen (paracetamol).
  * Antacids (e.g. TUMS, calcium carbonate, or magnesium hydroxide), proton pump inhibitors (e.g. omeprazole), H2 blockers (e.g. famotidine), or buffered vitamins.
* Epstein-Barr virus (EBV) negative nasopharyngeal carcinoma.

For Phase 2 only:

* Negative result on TrkA immunohistochemistry (IHC) assay.
* Have visceral crisis, defined as severe organ dysfunction and rapid progression of the cancer. (It is not about presence of visceral metastasis.)

For combination therapy with Pembrolizumab only:

* Serious adverse immune related adverse events (grade 3 or 4) with previous PD-1(L1) inhibitor therapy, that were symptomatic and required prolong immunosuppression (>6 weeks).
* Any grade Pneumonitis and Myocarditis related to prior PD-1(L1) inhibitor therapy.
* For subjects that received PD-1(L1) inhibitors before, there should be a washout period of at least 21 days between the last day of PD-1(L1) inhibitor and first day of study medications.
* Subjects who relapsed after prior treatment with PD-1(L1) inhibitors. Relapsed is defined as patients having best overall response of CR or PR after treatment with a PD-1(L1) inhibitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2018-06-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent Adverse Events (Phase 1) | First cycle (21 days per cycle)
  TEAE
To determine the recommended Phase 2 dose for VMD-928 (Phase 1) | First cycle (21 days per cycle)
  RP2D of monotherapy
To determine the RP2D of VMD-928 in combination with pembrolizumab (Phase 1) | First cycle (21 days per cycle)
  RP2D of combination therapy
Antitumor activity of VMD-928 in subjects with TrkA-driven tumors (Phase 2) | Up to 18 months
  Antitumor efficacy signal for monotherapy
Antitumor activity of VMD-928 in combination with pembrolizumab in subjects with TrkA-driven tumors (Phase 2) | Up to 18 months
  Antitumor efficacy signal for combination therapy

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of VMD-928. | On Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  AUC
Peak plasma concentration (Cmax) of VMD-928. | On Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  Cmax
Incidence of Dose Limiting Toxicities. | During the Cycle 1 (each cycle is 21 days)
  # of DLTs
Correlation between clinical antitumor and TrkA protein expression. | Up to the end of the Cycle 2 (each cycle is 21 days)
  Relationship of TrkA vs. efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Chair — VM Oncology
Locations (15):
- United States (14):
  - Providence Medical Foundation (site 209), Santa Rosa, California
  - Hartford Hospital (site 210), Hartford, Connecticut
  - The George Washington University Cancer Center (site 212), Washington D.C., District of Columbia
  - Holy Cross Hospital (site 213), Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Healthcare Systems (site 132), Pembroke Pines, Florida
  - Englewood Hospital and Medical Center (site 202), Englewood, New Jersey
  - Summit Medical Group (site 205), Florham Park, New Jersey
  - Atlantic Health System, Morristown Medical Center (site 124), Morristown, New Jersey
  - Presbyterian Kaseman Hospital (site 208), Albuquerque, New Mexico
  - Weill Cornell Medicine, Cornell University (site 126), New York, New York
  - Taylor Cancer Research Center (site 204), Maumee, Ohio
  - Cancer Care Associates of York (site 206), York, Pennsylvania
  - The University of Texas MD Anderson Cancer Center (site 127), Houston, Texas
  - Utah Cancer Specialists (site 203), Salt Lake City, Utah
- PanOncology Trials, Hospital Oncologico - Puerto Rico Medical Center, Río Piedras (site 200), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided